CLINICAL TRIAL: NCT04737616
Title: Continuous Monitoring and Management of Vaginal Health Via Multifunctional 1.7um Optical Coherence Tomography/Angiography Endoscopy
Brief Title: Continuous Monitoring and Management of Vaginal Health Via Multifunctional OCT/OCTA/OCE Endoscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Felicia Lane, Chair, Division of FPMRS, University of California, Irvine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20195446
Record Dates: First submitted 2021-01-22; First posted 2021-02-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: OCT: Optical coherence tomography; CO2: Carbon dioxide; GSM: genitourinary syndrome of menopause; OCE: Optical coherence angiography; OCTA:Optical coherence tomography with angiography
MeSH Terms: interventions — Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CO2 Laser +OCT (Experimental): Postmenopausal women with genitourinary syndrome of menopause who will receive CO2 vaginal laser treatment
  Interventions: Device: CO2 laser; Device: OCT
- OCT only (Experimental): Premenopausal, peri-menopausal and postmenopausal women who will only get one time OCT scan
  Interventions: Device: OCT

INTERVENTIONS:
Device: CO2 laser — Fractional CO2 vaginal laser for genitourinary syndrome of menopause
  Arms: CO2 Laser +OCT
Device: OCT — Optical coherence tomography endoscope

SUMMARY:
We have recently developed and optimized a vaginal Optical Coherence tomography/angiography endoscopy imaging system. This technology is able to obtain a comprehensive image of the vaginal epithelium, blood vessels, and lamina propria. The primary focus of this study is establishing the Optical Coherence Tomography system's capability of capturing vaginal changes that occur before and after menopause, as well as before and after treatment with fractional-CO2 laser therapy.

There are two aims of this study.

Aim 1:

1. To determine the feasibility and sensitivity of the integrated optical coherence endoscope to assess vaginal tissue integrity in pre, peri and postmenopausal women.

Aim 2:

To optically visualize the effects of fractional-CO2 laser treatment on vaginal tissue over the course of C02 vaginal laser therapy.

DETAILED DESCRIPTION:
The vaginal Optical Coherence tomography/angiography endoscopy imaging system. This technology is able to obtain a comprehensive image of the vaginal epithelium, blood vessels, and lamina propria. The primary focus of this study is establishing the Optical Coherence Tomography system's capability of capturing vaginal changes that occur before and after menopause, as well as before and after treatment with fractional-CO2 laser therapy.

There are two aims of this study.

Aim 1: To determine the feasibility and sensitivity of the integrated optical coherence endoscope to assess vaginal tissue integrity in pre, peri and postmenopausal women

We will enroll up to 90 women (age: 18 and older) who will be classified as pre-menopausal, peri- menopausal, or post-menopausal. There will be 30 women in each group. All enrolled subjects will first complete informed consents.

They will then fill out a questionnaire (the vulvovaginal symptom questionnaire) about their vaginal health. This will be followed by a pelvic exam to determine the vaginal health (vaginal health index) and to obtain a vaginal swab for assessment of the vaginal microbiome .

This will be followed by OCT scan of the vaginal tissue. There will be only one visit.

Aim 2: To optically visualize the effects of fractional-CO2 laser treatment on vaginal tissue over the course of C02 vaginal laser therapy.

Up to thirty Post-menopausal subjects with GSM who desire fractional-CO2 laser therapy, will be recruited.

Each visit will include: completion of a questionnaire (the vulvovaginal symptom questionnaire) about their vaginal health; followed by a pelvic exam to determine the vaginal health (vaginal health index) and to obtain a vaginal swab for assessment of the vaginal microbiome and an OCT scan of the vaginal tissue before the CO2 vaginal laser treatment.

This group will have a total of three visits with CO2 laser treatments. There will be a fourth visit which will include all the above study procedures except the CO2 laser treatment.

Subjects who complete 3 laser treatments will be offered participation in long term follow up with repeat OCT imaging every 3 months at 3, 6, 9 and 12 months after the final laser treatment to study the long- term effects of the laser treatment on the vaginal tissue.

ELIGIBILITY:
Inclusion criteria

Aim 1:

. Women who are premenopausal, peri-menopausal and postmenopausal

Aim 2:

. Postmenopausal women with genitourinary syndrome of menopause

Exclusion criteria

* history of pelvic irradiation
* Current pregnant or breastfeeding
* Use of hormone replacement therapy within three months of study enrollment
* Inability to read and understand english
* inability to follow research instructions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is for women only as it studies vaginal health.
Enrollment: 90 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Vaginal epithelial thickness (VET) | 2 years
  Vaginal epithelium thickness measured with the OCT.

SECONDARY OUTCOMES:
blood vessel density | 2 years
  The blood vessel density will be measured by OCT
Vaginal Health Index (VHI) | 2 years
  VHI to be measured on exam
Lactobacillus abundance | 2 years
  Lactobacillus abundance by RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Lane, MD, Principal Investigator — UC Irvine
Locations (1):
- Beckman Laser Institute and Medical Clinic, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No